CLINICAL TRIAL: NCT03694743
Title: Assessment of Postoperative Pain After Using 2Shape and Protaper Next Rotary Systems in Patients With Symptomatic Pulpitis in Mandibular Molars:A Randomized Clinical Trial
Brief Title: Post-operative Pain in 2Shape Versus Protaper Next Rotary Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ibrahim Mohamady, Ass.lecturer of endodotics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: dentistry cairo
Record Dates: First submitted 2018-09-29; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Pulpitis
Keywords: mandibular molars
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2Shape rotary system (Experimental): root canal preparation using 2Shape rotary system in mandibular molars with symptomatic pulpitis
  Interventions: Device: 2Shape rotary system
- Protaper Next rotary system (Active Comparator): root canal preparation using Protaper Next rotary system comparing to 2Shape rotary system in mandibular molars with symptomatic pulpitis
  Interventions: Device: 2Shape rotary system

INTERVENTIONS:
Device: 2Shape rotary system — root canal preparation

SUMMARY:
Pain after endodontic treatment is considered the most disturbing problem facing both the patient and the dentist especially in cases of symptomatic pulpitis as the patient is expecting to relief the pain that already exists.Therefore, this study aims to find a solution for the post-operative pain felt by the patient with symptomatic pulpitis in mandibular molars through comparing post-operative pain following use of 2Shape and Protaper Next rotary systems.

DETAILED DESCRIPTION:
Root canal preparation is the most important step in endodontic treatment. For successful treatment, pulp tissue, dentin debris and microorganisms should be completely eradicated from the root canal system.However, it has been reported that all the instrumentation techniques (manual or mechanical) cause debris extrusion into the periradicular tissue resulting in periapical inflammation that causes post-operative pain and flare up.

Instrumentation technique and instrument design were found to be related to the amount of debris extruded which is the main cause of post-operative pain. It has been reported that rotary NiTi systems cause less debris extrusion than manual instrumentation.

Within NiTi systems, instrument design, taper and tip size were found to affect debris extrusion. Therefore, new innovations in the instrument designs are introduced in order to reduce post-operative pain and flare up incidence.

Therefore, this study is established to compare the effect of 2 different rotary systems on postoperative pain in patients with symptomatic pulpitis.

The aim of the present study is to assess the effect of rotary instrumentation using Protaper Next rotary system versus 2Shape rotary system on postoperative pain and the number of analgesics taken by the patient following single visit root canal treatment in mandibular molars with symptomatic pulpitis.

Primary objective:

Comparing the intensity of post-operative pain using Numerical Rating Scale (NRS) immediately after root canal treatment and post-appointment at 6, 12, 24, 48 and 72hours.

Secondary objectives:

* The need for / and number of analgesic tablets taken within 3 days after end of endodontic treatment.
* Instrument separation during instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* - Medically free patients.
* Patients with symptomatic pulpitis in one of their mandibular molars.
* Patient's age ranges between 22 to 45 years with no sex predilection.
* Patients who can understand Numerical Analogue Scales (NRS).
* Patients able to sign informed consent.

Exclusion Criteria:

* - Patients having a systemic disorder.
* Presence of periapical lesion.
* Pregnant females.
* Patients who had taken analgesics during the last 12 hours preoperatively.
* Patients having active pain in more than one tooth.
* Non- educated patients.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
intensity of postoperative pain assessed by numerical rating scale Immediately after the end of treatment, and at 6, 12, 24, 48, and 72 hours. post-operative pain | 3 days
  using numerical rating scale ranges between (0-10) where 0 indicates no pain while 10 indicates maximum pain degree

SECONDARY OUTCOMES:
Need for / and number of analgesic tablets taken. | 3 days
  incidence and number of analgesic tablets will be recorded

OTHER OUTCOMES:
incidence of instrument seperation during endodontic treatment (instrument seperation means instrument fracture) | 1 day
  incidence will be recorded